CLINICAL TRIAL: NCT00730418
Title: A Prospective Study for the Effects of Chronic Use of Doxazosin on Alpha 1-adrenergic Receptors in Men With Benign Prostatic Hyperplasia
Brief Title: Effects of Chronic Use of Doxazosin in Men With Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Kyu-Sung Lee/Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2006-08-118
Record Dates: First submitted 2008-08-07; First posted 2008-08-08 (Estimated); Last update posted 2010-08-26 (Estimated); Status verified 2010-08

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; alpha Adrenergic Blockers; alpha-1 Adrenergic Receptor
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Doxazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- doxazosin 4mg (Experimental): doxazosin 4mg group
  Interventions: Drug: Doxazosin
- doxazosin 8mg (Experimental): doxazosin 8mg group
  Interventions: Drug: Doxazosin

INTERVENTIONS:
Drug: Doxazosin — Treatment with doxazosin 4mg daily for 24 mos
  Other Names: Cadura XL 4mg
  Arms: doxazosin 4mg
Drug: Doxazosin — Treatment with doxazosin 8mg daily for 24 mos
  Other Names: Cadura XL 8mg
  Arms: doxazosin 8mg

SUMMARY:
In this study, we investigate the changes of the expression of alpha adrenergic receptor in the prostate tissue during 2-yr medication period in the man with benign prostatic hyperplasia. And we also evaluate the efficacy and safety of 24 mo-treatment with doxazosin (4mg, 8mg)

DETAILED DESCRIPTION:
To compare the expression of alpha-1 adrenergic receptors, we will use various methodologies such as

* Real-time RT-PCR
* Radioligand receptor binding
* Western blot
* Immunohistochemistry

ELIGIBILITY:
Inclusion Criteria:

* 50 yrs or greater
* International prostatic symptom score >= 8
* Maximal flow rate < 15mL/sec
* baseline PSA 2.5-10 ng/mL
* Pathologically proven BPH
* No medication history for BPH
* Able to give fully informed consent

Exclusion Criteria:

* Previous use of alpha-blocker, 5-alpha reductase inhibitor
* Previous surgery for BPH
* Urologic cancer history
* Urethral stricture
* baseline PSA > 10ng/mL
* BP < 90/70 mmHg
* Orthotopic hypotension with syncope
* Serum Cr > 2.0 mg/dl, alanine aminotransferase > 1.5 times of normal limit
* Bacterial prostatitis within 1 year
* Urinary tract infection(UTI) more than 2 times within 1 year
* Active UTI or prostate biopsy within 1 month
* Unable to void
* Ped use because of incontinence
* Hypersensitivity to alpha-blocker that include quinazoline
* Unstable angina, Myocardial infarction, or cerebrovascular accident within 6 months
* Neurogenic bladder dysfunction (ex. multiple sclerosis, Parkinson's disease, Spinal injury etc.)
* Psychiatric problem
* Alcohol abuse or other drug abuse history
* Severe comorbidities unable to perform long-term trial
* seems not to be appropriate to this study because of any other reasons

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Expression of alpha-1 adrenoceptor | before treatment and 12mos and 24 mos after treatment

SECONDARY OUTCOMES:
International Prostate Symptom Score, Patient perception of bladder condition, Maximal flow rate of urine, Postvoid Residual, Prostate volume, Serum PSA level, Adverse events | before treatment and 3mos, 12mos, and 24mos after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kru-Sung Lee, Ph.D., M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea